CLINICAL TRIAL: NCT02141477
Title: A Phase II Study of Omacetaxine (OM) and Decitabine (DAC) in Older Patients With Acute Myelogenous Leukemia (AML) and High-Risk Myelodysplastic Syndrome (MDS)
Brief Title: Omacetaxine and Decitabine in Acute Myelogenous Leukemia (AML) and Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow Accrual-2 patients were registered Phase I and none in Phase II
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0812; NCI-2014-02157 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Leukemia
Keywords: Leukemia; Acute Myelogenous Leukemia; AML; High Risk Myelodysplastic Syndrome; MDS; Omacetaxine; Synribo; Homoharringtonine; Decitabine; Dacogen
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Homoharringtonine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Omacetaxine + Decitabine (Experimental): Phase I and Phase II Omacetaxine Dose: 1.25 mg/m2 subcutaneously every 12 hours on Days 1 - 3 of a 28 day cycle.
  Phase I Starting Decitabine Dose: 20 mg/m2 by vein on Days 1 - 5 of a 28 day cycle.
  Phase II Starting Decitabine Dose: Maximum tolerated dose from Phase I.
  Interventions: Drug: Omacetaxine; Drug: Decitabine

INTERVENTIONS:
Drug: Omacetaxine — Phase I and Phase II Omacetaxine Dose: 1.25 mg/m2 subcutaneously every 12 hours on Days 1 - 3 of a 28 day cycle.
  Other Names: Synribo; Homoharringtonine
Drug: Decitabine — Phase I Starting Decitabine Dose: 20 mg/m2 by vein on Days 1 - 5 of a 28 day cycle.
  Phase II Starting Decitabine Dose: Maximum tolerated dose from Phase I.
  Other Names: Dacogen

SUMMARY:
This clinical research study is made up of 2 phases. The goal of Phase 1 of the study is to test the safety of the combination of omacetaxine and decitabine and to find the best dose to give to future patients. The goal of Phase 2 of the study is to learn if this dose can help to control AML and/or MDS. The safety will then continue to be studied.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 2 groups of up to 6 participants (combined) will be enrolled in the Phase 1 portion of the study, and up to 60 participants will be enrolled in Phase 2.

If you are enrolled in Phase 1, the dose of decitabine you receive will depend on when you joined this study. If the first group of participants to receive decitabine has intolerable side effects, a second group will receive a lower dose.

If you are enrolled in Phase 2, you will receive decitabine at the highest dose that was tolerated in Phase 1.

All participants will receive the same dose level of omacetaxine.

Study Drug Administration:

Each cycle is 28 days.

Omacetaxine will be given as an injection under your skin 2 times each day, 12 hours apart (+/- 3 hours) on Days 1-3 of every cycle.

Decitabine will be given by vein over about 1 hour on Days 1-5 of every cycle.

Study Visits:

Every week (+/- 2 days), blood (about 2-3 teaspoons) will be collected for routine tests. If the disease appears to get better, this blood will only be drawn every 2-4 weeks while you are still receiving the study drugs, and every 4 to 8 weeks after that as long as you are on study. If you live far from the clinic, this blood and urine can be collected at a clinic close to your home, and the results will be reported to the study doctor.

At the beginning of every cycle, you will have a physical exam.

At Week 3 (+/- 7 days) and then every 4 weeks after that (+/- 7 days), you may (based on the results of your blood tests) have a bone marrow aspirate/biopsy collected to check the status of the disease and for cytogenetic testing.

Length of Study:

You may continue taking the study drugs for up to 3 years or as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

Follow Up:

You will have follow-up visits every 3-6 months for up to 5 years after you stop receiving the study drugs. At these visits, you will have a physical exam. If you cannot come to the clinic, you may just be called by the study staff and asked about your health. These calls should last about 5-10 minutes.

This is an investigational study. Omacetaxine is FDA approved and commercially available for the treatment of chronic myelogenous leukemia (CML). Its use in this study is investigational. Decitabine is FDA approved and commercially available for the treatment of MDS.

The study doctor can explain how the study drugs are designed to work.

Up to 66 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated AML (>/= 20% blasts) or AML M6. Patients with high-risk (intermediate-2 or high by IPSS or >/= 10% blasts) MDS will also be eligible. Prior therapy with hydroxyurea, biological or targeted therapy (e.g. flt3 inhibitors, other kinase inhibitors, azacitidine), or hematopoietic growth factors is allowed. No prior chemotherapy is allowed except for a single or a two day dose of cytarabine (up to 3 g/m2) for emergency use is also allowed as prior therapy.
2. Age >/= 70 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status </= 2.
4. Adequate hepatic (serum total bilirubin </= 1.5 x ULN, serum glutamate pyruvate transaminase (SGPT) and/or SGOT </= 2.5 x ULN) and renal function (creatinine </= 2.0 mg/dL).
5. Patients must be willing and able to review, understand, and provide written consent before starting therapy.
6. Men of childbearing potential who agree to use contraception prior to study entry and for the duration of participation.

Exclusion Criteria:

1. New York Heart Association (NYHA) class III or IV heart disease, active ischemia or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiac arrhythmia and requiring therapy, uncontrolled hypertension (blood pressure >/= 160 systolic and >/= 110 diastolic not responsive to antihypertensive medication), uncontrolled diabetes mellitus, or congestive heart failure.
2. Myocardial infarction in the previous 12 weeks (from the start of treatment).
3. Active and uncontrolled disease/infection as judged by the treating physician.
4. Acute promyelocytic leukemia (APL).

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
Safe Dose Combination of Omacetaxine (OM) and Decitabine (DAC) | 28 days
  Safe dose defined as highest dose level with </= 1 out of 6 patients experience a dose limiting toxicity (DLT) during first treatment cycle. DLT defined as clinically significant Grade 3 or 4 adverse event or abnormal laboratory value according to Common Toxicity Criteria for Adverse Effects (CTCAE) criteria assessed by treating physician as related to study drug (and unrelated to disease progression, intercurrent illness, or concomitant medications) occurring during the first 28 days on study.

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | 8 weeks
  Complete response rate (CRR) is defined as CR or CR with incomplete platelet recovery (CRp).

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org